CLINICAL TRIAL: NCT02242344
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Evaluation of the Safety, Efficacy and Pharmacokinetics of MICARDIS® (Telmisartan) in Children and Adolescents With Hypertension After Four Weeks of Treatment
Brief Title: Evaluation of the Safety, Efficacy and Pharmacokinetics of MICARDIS® (Telmisartan) in Children and Adolescents With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.403
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (3):
- telmisartan - low dose (Experimental)
  Interventions: Drug: Telmisartan
- telmisartan - high dose (Experimental)
  Interventions: Drug: Telmisartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: telmisartan - high dose; telmisartan - low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the blood pressure lowering effects of two doses of telmisartan over a four-week treatment period; to determine potentially effective doses for pediatric patients for future studies; to assess the safety and tolerability of two doses of telmisartan.

Pharmacokinetic objectives included the determination of the steady-state pharmacokinetics of telmisartan in children and adolescents aged 6 to <18 years, and to determine if age-related differences exist

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children and adolescents 6 to <18 years of age at time of informed consent/assent
2. Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local Institutional Review Boards (IRBs), and/or patient assent, when appropriate
3. Ability to stop any current antihypertensive therapy without unacceptable risk to the patient (Investigator's discretion)
4. Weight ≥20 kg and ≤120 kg
5. Hypertensive patients: in-clinic seated SBP ≥ 95th percentile based on age, height, and gender as defined in The Fourth Report on the Diagnosis, Evaluation and Treatment of High Blood Pressure in Children and Adolescents
6. Ability to swallow whole tablets

Exclusion Criteria:

1. Hypertension accompanied by symptoms or signs of central nervous system injury, including stroke, seizures, or encephalopathy, within 6 months prior to enrollment in the study
2. Children whose in-clinic seated BP measurements are 20 mmHg SBP or 10 mmHg DBP above the 95th percentile based on The Fourth Report on the Diagnosis, Evaluation and Treatment of High Blood Pressure in Children and Adolescents
3. Bilateral renal artery stenosis, unilateral renal artery stenosis in a solitary kidney, or uncorrected coarctation of the aorta
4. Congestive heart failure, valvular disease, or clinically significant cardiac rhythm disturbances
5. Bone marrow transplantation
6. Solid organ transplantation
7. Stroke
8. Chronic Kidney Disease with Glomerular Filtration Rate (GFR) to < 40 ml/min/1.73m2 by the Schwartz formula:

   Estimated GFR = (k x Height [cm]/ Serum Creatinine (mg/dL). k = 0.55 for all females and boys <13 years old; k = 0.7 in adolescent males ≥13 years old)
9. Clinically significant hepatic disease or abnormal liver function tests:

   1. Serum Glutamate-Oxaloacetate-Transaminase (Aspartate Aminotransferase) (SGOT), Serum Glutamate-Pyruvate-Transaminase (Alanine Aminotransferase) (SGPT), or Gamma-Glutamyl-Transferase (GGT) more than 2x upper limit of normal
   2. Total or direct bilirubin more than 1.5x upper limit of normal
10. Clinically significant gastrointestinal disease that may affect drug absorption or excretion (including gastroesophageal reflux, malabsorption, biliary disease, pancreatic disease)
11. Hyponatremia (serum sodium ≤130 mEq/L), hyperkalemia (Serum potassium ≥ 5.5 mEq/L), or other clinically significant electrolyte disorders
12. Significant hypoalbuminemia (serum albumin ≤2.5 g/dL)
13. Clinically significant neurological, psychiatric, pulmonary, hematological, or other condition that, in the opinion of the Investigator, will interfere with the safe and successful completion of the study
14. Hypersensitivity to angiotensin II receptor antagonists
15. Females who are of childbearing potential who:

    1. are pregnant/have a positive urine pregnancy test (UPT) prior to randomization (Visit 2), or
    2. are nursing, or lactating, or
    3. would not confirm abstinence (patients must be abstinent throughout the duration of the trial), or
    4. are not currently practicing one of the acceptable methods of birth control. Acceptable methods of birth control are limited to: Intra-Uterine Device (IUD), oral, implantable or injectable contraceptives and estrogen patch.
16. Concomitant therapy with any of the following agents:

    * Any angiotensin II receptor antagonist within four (4) weeks prior to randomization into the study
    * Any medication that could affect BP
    * Angiotensin Converting Enzyme (ACE) inhibitors within four (4) weeks prior to randomization into the study
    * Intravenous pulse steroid therapy within one month, daily treatment with oral corticosteroids ≥1 mg/kg/day)
    * Anticonvulsant medications
    * Bile acid binding agents
    * Any drug that may interfere with absorption of the study medication (e.g.antacids)
    * Drugs that may affect gastrointestinal motility (e.g. metoclopramide)
    * Cytotoxic agents within 12 months prior to enrollment into the study
17. Other investigational drugs or treatments within 30 days prior to enrollment
18. Patients who require two or more anti-hypertensive medications
19. Hereditary fructose intolerance
20. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated systolic blood pressure (SBP) | Baseline, after 4 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in seated diastolic blood pressure (DBP) | Baseline, after 4 weeks of treatment
Response rate of blood pressure | after 4 weeks
  defined as both SBP and DBP < 95th percentile at the patient's final visit based on age, height, and gender
Cmax,ss (maximum concentration of the analyte in plasma at steady state over a uniform dosing interval) | 72 hours after last study drug administration
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval) | 72 hours after last study drug administration
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | 72 hours after last study drug administration
Cavg (Average concentration of the analyte in plasma at steady state) | 72 hours after last study drug administration
tmax,ss (time from dosing to maximum concentration at steady state) | 72 hours after last study drug administration
AUCτ,ss (area under the concentration time curve of the analyte in plasma at steady state over a uniform dosing interval) | 72 hours after last study drug administration
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | 72 hours after last study drug administration
MRTpo,ss (mean residence time of the analyte in the body at steady state) | 72 hours after last study drug administration
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | 72 hours after last study drug administration
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) | 72 hours after last study drug administration
PTF (peak trough fluctuation) | 72 hours after last study drug administration
Number of patients with adverse events | up to 45 days

REFERENCES:
- See also: Related Info — http://journals.sagepub.com/doi/abs/10.1177/0009922810363609